CLINICAL TRIAL: NCT02870218
Title: Abuse Liability of Reduced Nicotine Content Cigarettes in the Context of Concurrent E-Cigarette Use
Acronym: DUAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jed Rose, President and CEO, Rose Research Center, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201602820; GRANT12052089 (Other: Grants.gov); 5R01DA042541-03 (NIH)
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Nicotine Addiction; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- 0.40mg Nicotine Cigarette w/ e-Cigarette (Active Comparator): Participants will be assigned to smoke 0.40mg nicotine Spectrum cigarettes for 12 weeks with unlimited access to JUUL e-cigarettes.
  Smoking research cigarettes with e-cigarette
  Interventions: Drug: Smoking research cigarettes with e-cigarette
- 1.40mg Nicotine Cigarette w/ e-Cigarette (Active Comparator): Participants will be assigned to smoke 1.40mg nicotine Spectrum cigarettes for 12 weeks with unlimited access to JUUL e-cigarettes.
  Smoking research cigarettes with e-cigarette
  Interventions: Drug: Smoking research cigarettes with e-cigarette
- 2.50mg Nicotine Cigarette w/ e-Cigarette (Active Comparator): Participants will be assigned to smoke 2.50mg nicotine Spectrum cigarettes for 12 weeks with unlimited access to JUUL e-cigarettes.
  Smoking research cigarettes with e-cigarette
  Interventions: Drug: Smoking research cigarettes with e-cigarette
- 5.60mg Nicotine Cigarette w/ e-Cigarette (Active Comparator): Participants will be assigned to smoke 5.60mg nicotine Spectrum cigarettes for 12 weeks with unlimited access to JUUL e-cigarettes.
  Smoking research cigarettes with e-cigarette
  Interventions: Drug: Smoking research cigarettes with e-cigarette
- 16.9mg Nicotine Cigarette w/ e-Cigarette (Active Comparator): Participants will be assigned to smoke 16.9mg nicotine Spectrum cigarettes for 12 weeks with unlimited access to JUUL e-cigarettes.
  Smoking research cigarettes with e-cigarette
  Interventions: Drug: Smoking research cigarettes with e-cigarette
- Halo G6 & Tribeca e-liquid (Experimental): Difference detection assessments.
  Nicotine discrimination thresholds
  Interventions: Drug: Nicotine discrimination thresholds
- Spectrum Research Cigarette (Experimental): Difference detection assessments.
  Nicotine discrimination thresholds
  Interventions: Drug: Nicotine discrimination thresholds

INTERVENTIONS:
Drug: Smoking research cigarettes with e-cigarette — Smoking research cigarettes with varying levels of nicotine with unlimited access to 15 mg/ml nicotine-containing e-cigarettes.
  Other Names: Spectrum Cigarettes; JUUL e-Cigarette
  Arms: 0.40mg Nicotine Cigarette w/ e-Cigarette; 1.40mg Nicotine Cigarette w/ e-Cigarette; 16.9mg Nicotine Cigarette w/ e-Cigarette; 2.50mg Nicotine Cigarette w/ e-Cigarette; 5.60mg Nicotine Cigarette w/ e-Cigarette
Drug: Nicotine discrimination thresholds — Measure of nicotine thresholds for detecting and recognizing the addictive, rewarding effects of smoking.
  Other Names: Halo G6 with Tribeca e-liquid
  Arms: Halo G6 & Tribeca e-liquid; Spectrum Research Cigarette

SUMMARY:
Three hundred-twenty (320) adult smokers of menthol or non-menthol combustible cigarettes will be recruited and randomly assigned to one of five groups (n=64/group), who will be asked to switch for 12 weeks to ad libitum use of combustible cigarettes (matched to subjects' menthol preference) containing either 0.4, 1.4, 2.5, 5.6 or 16.9 mg nicotine (standardized nicotine yields ranging from 0.02-0.80 mg/cigarette), respectively. Each group will include 32 heavy (≥ 20 cigarettes/day), and 32 light smokers (≤10 cigarettes/day), who are hypothesized to be more sensitive to nicotine's reinforcing effects. Participants will also have free access to nicotine-containing e-cigarettes (JUUL) throughout the 12-week period. Abuse liability of combustible cigarettes will be assessed by behavioral (cigarettes/day, time to first cigarettes), self-report (rewarding effects, withdrawal symptoms) and biochemical indices (expired air carbon monoxide, cotinine blood sampling).

In laboratory sessions, we will measure nicotine thresholds for detecting and recognizing the addictive, rewarding effects of smoking. This study is designed to help the FDA identify a target nicotine threshold that will not attract young people to smoking or induce relapse in former smokers. Additionally, we will determine the level of cigarette nicotine reduction that will be tolerated without inducing dissatisfaction in smokers, information that is relevant to the FDA for designing a stepwise nicotine reduction policy that can be implemented without widespread objections. The knowledge gained from this project will greatly increase our knowledge of nicotine addiction and will help frame an FDA policy relating to the regulation of the nicotine content of tobacco. Ultimately, a well-designed nicotine reduction policy has the potential to greatly reduce the enormous toll of death and disease caused by cigarette smoking.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is healthy as judged by the Investigator based on all available assessments from the Screening Period (e.g., safety laboratory, vital signs, physical examination, ECG, concomitant medications and medical history).
2. Subject smokes on average four days a week for the last 12 months.
3. Subject has no intention of quitting smoking within the next 90 days.
4. Owns a smart phone with text message and data capabilities.
5. Willingness to use and ability to operate e-cigarettes.
6. Willingness to smoke Research Cigarettes.

Exclusion Criteria:

1. Any medical or psychiatric condition (or associated symptoms or medications) determined by a medical professional to be severe enough to be disruptive to the study.
2. Severe or uncontrolled psychiatric disease with the exception of anxiety disorders, obsessive-compulsive disorder (OCD) and attention deficit hyperactivity disorder (ADHD);
3. Pregnant or nursing (by self-report) or positive pregnancy test;
4. Daily use of:

   1. Experimental (investigational) drugs that are unknown to subject;
   2. Smokeless tobacco (chewing tobacco, snuff), cigars, pipes and hookah;
   3. e-cigarettes;
5. Use in the past 30 days of nicotine replacement therapy or other smoking cessation product
6. Positive drug screen for cocaine

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Expired air CO Measurement | 12 Weeks
  To determine the effects of cigarette nicotine content manipulations on abuse liability as measured by exhaled breath CO.

SECONDARY OUTCOMES:
Nicotine discrimination tests to determine nicotine detection thresholds | Weeks 1, 2,8,10,12 and 14
  Results of the laboratory discrimination tests will be analyzed descriptively to determine nicotine detection thresholds. Thresholds will be calculated based on both group-averaged data as well as by using the best estimates of individual thresholds calculated from each smoker's data. Group averaged data will be determined by graphically plotting the overall percent correct against nicotine concentration.
Nicotine discrimination tests to determine nicotine recognition thresholds | Weeks 1, 2,8,10,12 and 14
  Results of the laboratory discrimination tests will be analyzed descriptively to determine nicotine recognition thresholds. Thresholds will be calculated based on both group-averaged data as well as by using the best estimates of individual thresholds calculated from each smoker's data. Group averaged data will be determined by graphically plotting the overall percent correct against nicotine concentration.
Extent of e-cigarette use based on self-report | 12 Weeks
  To determine whether the abuse liability of combustible cigarettes is related to the nicotine intake from e-cigarettes or to total nicotine intake, regression analyses will be conducted to correlate indices of abuse liability to levels of cotinine as well as to the estimated intake of nicotine from cigarettes and e-cigarettes based on self-reported values.
Extent of e-cigarette use based on self-report cotinine levels | 12 Weeks
  To determine whether the abuse liability of combustible cigarettes is related to the nicotine intake from e-cigarettes or to total nicotine intake, regression analyses will be conducted to correlate indices of abuse liability to levels of cotinine as well as to the estimated intake of nicotine from cigarettes and e-cigarettes.
Mean number of research cigarettes smoked per day as primary index of abuse liability | 12 Weeks
  To assess the effects of cigarette nicotine content on abuse liability among smokers who also use e-cigarettes. The primary index of abuse liability will be mean number of research cigarettes smoked per day. Secondary outcome measures comprise expired air carbon monoxide (CO), Fagerström Test for Nicotine Dependence (FTND) score, withdrawal symptoms and cognitive performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Rose Research Center, LLC
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No